CLINICAL TRIAL: NCT02142751
Title: Phase 3, Randomized, Controlled Multicentric, Open-label Clinical Trial to Prove Non-Inferiority of Fosfomycin vs Meropenem or Ceftriaxone in the Treatment of Bacteriemic Urinary Infection Due to Multidrug Resistance in E.Coli
Brief Title: Fosfomycin Versus Meropenem or Ceftriaxone in Bacteriemic Infections Caused by Multidrug Resistance in E.Coli
Acronym: FOREST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Spanish Network for Research in Infectious Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FOREST
Record Dates: First submitted 2014-05-13; First posted 2014-05-20 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Infection Due to ESBL Escherichia Coli
Keywords: Escherichia coli; Extended-spectrum β-lactamases (ESBLs); Bacteremia; Urinary tract infection; Bloodstream infection; Fosfomycin; Meropenem; Pharmacokinetics; intestinal colonization; Recurrence; multidrug resistance E.coli; Ceftriaxone
MeSH Terms: conditions — Escherichia coli Infections; Bacteremia; Urinary Tract Infections; Sepsis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Fosfomycin sodium intravenous (Experimental): 4g every 6 hours iv (60 min infusion)
  Interventions: Drug: Fosfomycin sodium intravenous
- Meropenem intravenous (Active Comparator): 1g every 8 hours (15-30 min infusion)
  Interventions: Drug: Meropenem intravenous
- Ceftriaxone intravenous (Other): 1g every 24h (2-4 min)
  Interventions: Drug: Ceftriaxone intravenous

INTERVENTIONS:
Drug: Fosfomycin sodium intravenous — 4g every 6 hours iv (60 min infusion)
  Other Names: Generic name: Fosfomycin; Pharmaceutical form: solution for infusion; ATC code: J01J3
  Arms: Fosfomycin sodium intravenous
Drug: Meropenem intravenous — 1g every 8 hours (15-30 min infusion) It depends on strain sensitivity: Strain with resistance to cephalosporins
  Other Names: Generic name: Meropenem; Pharmaceutical form: solution for infusion; ATC code: J01D5
  Arms: Meropenem intravenous
Drug: Ceftriaxone intravenous — 1g every 24 hours iv (2-4 min infusion) It depends on strain sensitivity: Strain with resistance to quinolone but sensitivity to cephalosporins
  Other Names: generic name: ceftriaxone; Pharmaceutical form: solution for infusion; ATC code:J01DA
  Arms: Ceftriaxone intravenous

SUMMARY:
Enterobacterieaceae (and specially Escherichia coli) showing resistance due to multidrug-resistant Escherichia coli, plasmid mediated AmpC or quinolone resistance caused by chromosomal mechanisms have spread worldwide during the last decades. This is important because many of these isolates are also resistant to other first-line agents such as fluoroquinolones or aminoglycosides, leaving few available options for therapy, and this condition is associated with increased morbidity- mortality and length of hospital stay. While carbapenems are considered the drugs of choice for multidrug-resistant Escherichia coli and AmpC producers, recent data suggests that certain alternatives may be suitable for some types of infections.

At the present time, finding therapeutic alternatives to carbapenems and cephalosporins for the treatment of invasive infections due to multidrug-resistant Escherichia coli is critical. Fosfomycin was discovered more than 40 years ago but was not investigated according to present standards, and thus is not used in clinical practice except in desperate situations. It is one of the so-considered neglected antibiotics with high potential interest for the future.

With the aim of demonstrate the clinical non-inferiority of intravenous fosfomycin compared to meropenem or ceftriaxone in the treatment of bacteraemic urinary tract infections caused by multidrug-resistant Escherichia coli . The investigators propose a "real practise" randomised, controlled, multicentre phase III clinical trial to compare the clinical and microbiological efficacy and safety of intravenous fosfomycin (4 grammes every 6 hours) with meropenem (1 gramme every 8 hours) or ceftriaxone (1 gramme every 24 hours) as targeted therapy of the previously specified infection; change to oral therapy according to predefined options is allowed in both arms after 5 days. Follow-up for the study is planned up to 60 days.

DETAILED DESCRIPTION:
The FOREST study is a phase 3, randomised, controlled, multicentric, open-label clinical trial to prove the noninferiority of fosfomycin versus meropenem in the targeted treatment of bacteraemic UTI due to ESBL-EC, designed as a real practice trial. It is a non-commercial, investigator-driven clinical study funded through a public competitive call by Instituto de Salud Carlos III, Spanish Ministry of Economy (PI13/01282).

The study is coordinated by investigators from Hospital Universitario Virgen Macarena in Seville, Spain; the sponsorship is performed by Fundación Pública Andaluza para la Gestión de la Investigación en Salud de Sevilla (FISEVI), of which the sponsor-scientific responsibilities are delegated to the CTU (Clinical Trial Unit-Hospital Universitario Virgen del Rocío, Seville, Spain). All participating patients or their relatives must give written informed consent before any study procedures occur, including the withdrawal of biological samples for the study.

The hypothesis to test is that intravenous fosfomycin is not inferior to meropenem for the targeted treatment of bacteraemic UTI caused by ESBL-EC in terms of efficacy.

The primary objective of the study is to demonstrate that intravenous fosfomycin is not inferior to meropenem for reaching clinical and microbiological cure 5-7 days after the completion of treatment.

Secondary objectives include comparing the early clinical and microbiological response, 30-day mortality, hospital stay, recurrence rate, safety and impact on intestinal colonisation by MDR Gram-negative bacilli, evaluation of the rate of resistance development to fosfomycin and blood level concentration of fosfomycin.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old hospitalized patients
* Negative pregnancy test in fertile women
* Episode of clinically-significant monomicrobial urinary BSI due to multidrug-resistant E.coli susceptible to fosfomycin and meropenem or ceftriaxone
* Urinary sepsis with multidrug resistant E. coli isolation from the blood cultures, requires at least one clinical criteria and one of the following urinalysis criteria:

Clinical criteria

* UTI symptoms (dysuriac, urgency, suprapubic pain or pollakiuria)
* Lumbar back pain
* Cost-vertebral angle tenderness
* Altered mental status in people up to 70 years old
* Intermittent or permanent indwelling foley catheter (or withdrawal during 24 hours previous) even without urinary symptoms urinalysis criteria
* Urine dipstick test positive for either nitrites or leukocyte esterase
* Positive urine culture - Signed informed consent form (ICF) executed prior to protocol screening assessments

Exclusion Criteria:

* Polymicrobial bacteremia
* No drainage of renal abscess or obstructive uropathy unresolved
* Pregnant or careening women
* Haematogenous infection
* Other concomitant infection
* Renal transplantation recipients
* Polycystic kidney
* Hypersensitivity and/or intolerance to meropenem or fosfomycin or ceftriaxone
* Palliative care or life expectance < 90 days
* Septic shock at time of randomization
* New York Heart Association (NYHA) functional Class IV, hepatic cirrhosis or renal impairment receiving dialysis
* Active empiric treatment >72 hours
* Late randomization >24 hours after multidrug resistant.coli blood culture´s identification
* Participation in other clinical trial with active treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Clinical and microbiological cure rate | Day 5-7 after end of treatment (test of cure)
  Clinical Cure: Complete resolution of infection symptoms (bacteremia and/or urinary tract infection-UTI-), present at the day on which blood culture was drawn.
  Microbiological cure: Negative blood culture at day 5-7 after end of treatment. Besides this, if UTI was confirmed with a positive urine culture with the same microorganism than the blood culture, this culture should become negative.

SECONDARY OUTCOMES:
Early clinical response | After 5 -7 days of complete treatment (from the first day of study drugs administration)
  The infection was completely resolved after 5-7 days of complete treatment
Mortality | At day 30 of follow-up
  Death for any reason.
Length of hospital stay | At day 30 of follow-up
  It is defined as the time from admission to hospital discharge
Safety of intravenous fosfomycin in this indication | To the last visit, at 60 plus-minus 10 days (from the first day of study drugs administration)
  Gathering any related adverse event from the informed consent form signature to the end of follow-up.
Recurrences (relapse and reinfection) rate | To the last visit, at 60 plus-minus 10 days (from the first day of study drugs administration)
  Relapse: new symptoms of UTI in patient with previously considered as clinical or microbiological cured in the visit of day 5-7 plus positive urine or blood cultures with the same microorganism isolated than the initial culture.
  Re-infection: same definition but with different strain in the culture results.
Fosfomycin steady-state plasma concentration | At 3 days after treatment started
  Therapeutic drug monitoring of fosfomycin, basic pharmacokinetic parameters will be determined.
Microbiota impact of study treatment bacilli | Screening, day 5-7, day 12
  Study treatment impact in the gut colonization of MDRGNB (Multi drug resistant Gram negative bacilli)
Emergence of resistant clinical isolates of Escherichia coli to fosfomycin and meropenem | participants will be followed for the duration of fosfomycin, an expected average of 14 days
  Frequency of strains that develop resistance and detection of resistance mechanisms in fosfomycin treatment arm.
Early microbiological response | within the first 5 days after treatment started
  Cultures are negative
Safety of intravenous antibiotic administration in this indication | To the last visit, at 60 plus-minus 10 days (from the first day of study drugs administration)
  Gathering any related adverse event from the informed consent form signature to the end of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: JESUS RODRIGUEZ-BAÑO, MD, PhD, Study Chair — Spanish Network for Research in Infectious Diseases
Locations (22):
- Spain (22):
  - Hospital Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria, Gran Canarias
  - Hospital Arnau de Vilanova, Vilanova, Lleida
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Marina Baixa, Alicante
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Parc Salud Mar, Barcelona
  - Hospital de la Santa Creu i San Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital de Cruces, Bilbao
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Royo Villanova, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sojo-Dorado J, Lopez-Hernandez I, Rosso-Fernandez C, Morales IM, Palacios-Baena ZR, Hernandez-Torres A, Merino de Lucas E, Escola-Verge L, Bereciartua E, Garcia-Vazquez E, Pintado V, Boix-Palop L, Natera-Kindelan C, Sorli L, Borrell N, Giner-Oncina L, Amador-Prous C, Shaw E, Jover-Saenz A, Molina J, Martinez-Alvarez RM, Duenas CJ, Calvo-Montes J, Silva JT, Cardenes MA, Lecuona M, Pomar V, Valiente de Santis L, Yague-Guirao G, Lobo-Acosta MA, Merino-Bohorquez V, Pascual A, Rodriguez-Bano J; REIPI-GEIRAS-FOREST group. Effectiveness of Fosfomycin for the Treatment of Multidrug-Resistant Escherichia coli Bacteremic Urinary Tract Infections: A Randomized Clinical Trial. JAMA Netw Open. 2022 Jan 4;5(1):e2137277. doi: 10.1001/jamanetworkopen.2021.37277. PMID 35024838
- [Derived] Rosso-Fernandez C, Sojo-Dorado J, Barriga A, Lavin-Alconero L, Palacios Z, Lopez-Hernandez I, Merino V, Camean M, Pascual A, Rodriguez-Bano J; FOREST Study Group. Fosfomycin versus meropenem in bacteraemic urinary tract infections caused by extended-spectrum beta-lactamase-producing Escherichia coli (FOREST): study protocol for an investigator-driven randomised controlled trial. BMJ Open. 2015 Mar 31;5(3):e007363. doi: 10.1136/bmjopen-2014-007363. PMID 25829373
- See also: Spanish Network Research in Infectious Diseases (Red Española de Investigación en Patología Infecciosa [REIPI]) — http://www.reipi.org/